CLINICAL TRIAL: NCT00427999
Title: A Single Stage Phase II, Multi-centre, Open Label Study of Imatinib in Combination With Pioglitazone, Etoricoxib, Dexamethasone and Low-dose Treosulfane for Anti-inflammatory and Angiostatic Treatment in Patients With Hormone-refractory Prostate Cancer
Brief Title: Combined Antiinflammatory and Angiostatic Therapy in Patients With Hormone-refractory Prostate Cancer
Acronym: INV342
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE59; 2006-000218-19
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: Hormone-refractory; prostate cancer; multitargeted; tyrosinkinase
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Imatinib Mesylate; treosulfan; Etoricoxib; Pioglitazone; Dexamethasone; dexamethasone acetate

ARMS (1):
- STI571+ pioglitazone+ etoricoxib + dexamethasone + treosulfane (Experimental): STI571 (imatinib) 400mg po daily + pioglitazone 60mg po daily + etoricoxib 60mg po daily + dexamethasone 1mg po daily + treosulfane 500mg po daily for 24 weeks
  Interventions: Drug: imatinib mesylate; Drug: Treosulfane; Drug: etoricoxib; Drug: pioglitazone; Drug: dexamethasone

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: Gleevec; Glivec
Drug: Treosulfane
  Other Names: Ovastat
Drug: etoricoxib
  Other Names: Arcoxia
Drug: pioglitazone
  Other Names: Actos
Drug: dexamethasone
  Other Names: Fortecortin

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability and safety of a multi-targeted therapy in patients with hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed prostate carcinoma, which has proven progression after primary hormone therapy (surgical or medicinal castration).
* Patients must have increasing PSA levels (within 3 months prior to enrollment) with at least two consecutively increasing PSA levels.
* PSA value before inclusion must be at least 5 ng/ml
* At least 18 years of age.
* At least capable of self care and up of at least 50% of waking hours (ECOG performance status 0 - 2), adequate bone marrow function and lab results.

Exclusion criteria:

* Change of hormone therapy within 6 weeks prior inclusion
* Prior chemotherapy
* Therapy with Imatinib, or therapy with other inhibitors of tyrosinkinase.
* Second neoplasm diagnosed within 5 years before study start.
* Patients who require therapy with warfarin
* Known diagnosis of HIV, hepatitis B, or hepatitis C infection.
* Severe, unstable, or uncontrolled medical disease which would confound diagnoses or evaluations required by the protocol, including severe cardiac insufficiency
* Surgical therapy within 4 weeks before inclusion.
* Prior therapy with isotopes strontium or rhenium.
* Radiation therapy to > 25% of bone marrow within 4 weeks before inclusion.
* Treatment with other experimental substances within 30 days before study start.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (9):
- Germany (9):
  - Novartis Investigative Site, Bad Reichenhall
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Passau
  - Novartis Investigative Site, Planegg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 15 centers 72 patients were screened, 67 enrolled, of which 65 were treated and 33 completed the treatment phase. Intent to Treat (ITT) population included 61 patients. For the extension follow-up phase 19 patients were included in the safety analysis.
Period: Overall Study
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Started | 65
Intent to Treat (ITT) | 61
Extension Follow-up | 19
Completed | 33
Not Completed | 32
Not completed — Adverse Event | 6
Not completed — Abnormal laboratory values | 1
Not completed — Unsatisfactory therapeutic effect | 13
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 9
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 65

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: To investigate the effect of a treatment with Imatinib mesylate, Pioglitazone , Etoricoxib, and Dexamethasone in combination with metronomic chemotherapy (Treosulfane) on the PSA response rate in patients with hormone refractory prostate cancer. A patient will be defined as a responder if a PSA decline of at least 50%, which must be confirmed by a second PSA value 4 weeks later, is observed. A patient will be defined as a non-responder if PSA has not decreased during treatment. Non-response is defined as a 25% increase over the baseline on-study which is confirmed (equal or more) by a second value 4 weeks apart. The absolute increase must account for > 5 ng/ml.
Time Frame: up to 24 weeks
Population: Intent to Treat (ITT) includes the 61 patients treated.
Measure: Number; unit: participants
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 61
participants
  PSA responder - No | 38
  PSA responder - Yes | 23

2. Secondary Outcome: Time to PSA Response
Description: Time to PSA response, defined as the time from first administration of study drugs to the first PSA value of a confirmed PSA response. Non-responders will be censored with date of final visit/premature discontinuation for the analysis. Median time to PSA response was not achieved
Time Frame: every 4 weeks up to 24 weeks
Population: Intent to Treat (ITT) includes the 61 patients treated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 61
days | NA [NA to NA] — Median time to PSA response was not achieved

3. Secondary Outcome: Time to Progression-free Survival
Description: Progression-free survival, defined as the time from first administration of study drugs to the first PSA value of a PSA non-responder. Responders will be censored with date of PSA response for the analysis. The median time to PSA progression free survival was not achieved
Time Frame: every 4 weeks up to 24 weeks
Population: Intent to Treat (ITT) includes the 61 patients treated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 61
days | NA [NA to NA] — The median time to PSA progression free survival was not achieved

4. Secondary Outcome: Overall Survival Rate
Description: Overall survival (OS) is defined as time from randomization to death from any cause or last date known alive. The median time to overall survival rate was not achieved
Time Frame: every 4 weeks up to 24 weeks
Population: Intent to Treat (ITT) includes the 61 patients treated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 61
days | NA [NA to NA] — The median time to overall survival rate was not achieved

5. Secondary Outcome: Quality of Life Assessed With EORTC-30
Description: Health-related quality of life was assessed with the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-30) questionnaire and was presented descriptively. The EORTC QLQ-C30 is a questionnaire including following sub-scales: global health status, functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social activity), symptom scales (fatigue, nausea and vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties). Scores are averaged for each scale and transformed to 0-100 scale; higher score indicates better quality of life on global health status and functional scales and worse quality of life on symptom scales and financial difficulty scale.
Time Frame: baseline and Final Visit (week 24)
Population: Intent to Treat (ITT) includes the 61 patients treated
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | STI571+ Pioglitazone+ Etoricoxib + Dexamethasone + Treosulfane
Number analyzed (Participants) | 61
scores on a scale
  Baseline: financial difficulties (n=49) | 11.6 (16.03)
  Baseline: appetite loss (n=50) | 16.0 (29.54)
  Baseline: dyspnea (n=49) | 20.4 (27.06)
  Baseline: constipation (n=50) | 14.0 (28.64)
  Baseline: role functioning (n=50) | 74.0 (28.80)
  Baseline: insomnia (n=49) | 34.0 (34.35)
  Baseline: cognitive functioning (n=49) | 87.1 (16.41)
  Baseline: diarrhea (n=50) | 9.3 (21.34)
  Baseline: physical functioning (n=50) | 81.7 (17.19)
  Baseline: pain (n=50) | 32.3 (32.89)
  Baseline: emotional functioning (n=49) | 64.6 (21.89)
  Baseline: social functioning (n=49) | 72.4 (26.69)
  Baseline: fatigue (n=50) | 32.9 (26.08)
  Baseline: global health status (n=49) | 60.0 (18.24)
  Baseline: nausea & vomiting (n=50) | 26.0 (28.80)
  Final Visit: financial difficulties (n=42) | 19.0 (28.65)
  Final Visit: appetite loss (n=43) | 24.0 (33.59)
  Final Visit: dyspnea (n=43) | 38.8 (29.03)
  Final Visit: constipation (n=43) | 6.2 (15.01)
  Final Visit: role functioning (n=43) | 55.4 (31.01)
  Final Visit: insomnia (n=42) | 31.7 (32.05)
  Final Visit: cognitive functioning (n=43) | 81.8 (20.51)
  Final Visit: diarrhea (n=43) | 13.2 (23.16)
  Final Visit: physical functioning (n=43) | 66.7 (25.32)
  Final Visit: pain (n=43) | 26.0 (30.06)
  Final Visit: emotional functioning (n=43) | 61.8 (28.42)
  Final Visit: social functioning (n=43) | 64.0 (32.52)
  Final Visit: fatigue (n=43) | 46.0 (29.05)
  Final Visit: global health status (n=43) | 51.0 (21.76)
  Final Visit: nausea & vomiting (n=43) | 44.6 (31.01)

ADVERSE EVENTS:
Description: In 15 centers 72 patients were screened, 67 enrolled, of which 65 were treated and 33 completed the treatment phase. Intent to Treat (ITT) population included 61 patients. For the extension follow-up phase 19 patients were included in the safety analysis.
Groups:
- STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Core): STI571 (imatinib) 400mg po daily + pioglitazone 60mg po daily + etoricoxib 60mg po daily + dexamethasone 1mg po daily + treosulfane 500mg po daily for 24 weeks (Core)
- STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Ext): Extension follow-up
Arm/Group | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Core) | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Ext)
Serious Adverse Events (participants affected / at risk) | 22/65 | 7/19
Other Adverse Events (participants affected / at risk) | 65/65 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Core) (N=65) | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Ext) (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 1
Disease progression (General disorders) | 1 | 1
Drug ineffective (General disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Postrenal failure (Renal and urinary disorders) | 2 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Core) (N=65) | STI571+Pioglitazone+Etoricoxib+Dexamethasone+Treosulfane(Ext) (N=19)
Anaemia (Blood and lymphatic system disorders) | 21 | 7
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 19 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 4 | 0
Vertigo (Ear and labyrinth disorders) | 7 | 3
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Cushing's syndrome (Endocrine disorders) | 11 | 1
Cushingoid (Endocrine disorders) | 4 | 3
Hypogonadism male (Endocrine disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 5 | 2
Lacrimation increased (Eye disorders) | 8 | 0
Visual acuity reduced (Eye disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 27 | 6
Gastric polyps (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 28 | 5
Toothache (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 16 | 3
Asthenia (General disorders) | 7 | 1
Face oedema (General disorders) | 15 | 4
Fatigue (General disorders) | 21 | 9
General physical health deterioration (General disorders) | 1 | 3
Generalised oedema (General disorders) | 1 | 2
Inflammation (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 1
Necrosis (General disorders) | 0 | 1
Oedema (General disorders) | 24 | 6
Oedema peripheral (General disorders) | 35 | 12
Pain (General disorders) | 5 | 0
Pyrexia (General disorders) | 2 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Gingivitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 7 | 3
Otitis media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0
Blood albumin decreased (Investigations) | 3 | 2
Blood alkaline phosphatase increased (Investigations) | 7 | 1
Blood creatinine increased (Investigations) | 9 | 5
Blood fibrinogen increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 10 | 4
Blood potassium decreased (Investigations) | 2 | 1
C-reactive protein increased (Investigations) | 4 | 3
Haematocrit decreased (Investigations) | 2 | 2
Lymphocyte count decreased (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
Occult blood (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Prostatic specific antigen increased (Investigations) | 2 | 2
Protein total decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 1 | 2
Reticulocyte count increased (Investigations) | 0 | 1
Weight increased (Investigations) | 13 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 1
Zinc deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 6 | 0
Dysgeusia (Nervous system disorders) | 7 | 1
Headache (Nervous system disorders) | 11 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 2
Polyneuropathy (Nervous system disorders) | 7 | 6
Depression (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Sleep disorder (Psychiatric disorders) | 6 | 3
Kidney fibrosis (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Renal pain (Renal and urinary disorders) | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Skin dystrophy (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Extravasation blood (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 5 | 0
Lymphoedema (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.